CLINICAL TRIAL: NCT02135172
Title: Does Breaking Sedentary Time Improve Glucose Regulation in Women With Impaired Glucose Tolerance? A Balanced Incomplete Block Design Study
Brief Title: Breaks in Sedentary Time and Glucose Regulation in Women
Acronym: ACUTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 0376
Record Dates: First submitted 2014-01-02; First posted 2014-05-09 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance | interventions — Sitting Position; Standing Position; Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sitting (Experimental): During the sitting treatment condition, walking and standing will be restricted. Participants will be in a designated room with access to a computer, books/magazines throughout the day. Participants will have a cannula fitted and the first of the half-hourly blood samples will be taken (time point: -1hr). Participants will then be asked to sit quietly for 60 minutes to achieve a steady state. Following this, participants will have another blood sample taken and then be provided with a standardised mixed meal breakfast (09:00am) (time point: 0h). Blood sampling will continue at 30 minutes intervals for 3 hours following breakfast. A second, lunch meal (12:00pm), will be then be consumed over 15 minutes. Blood sampling will then continue at 30 minute intervals for 3 hours following lunch.
  Interventions: Behavioral: Sitting
- Standing (Experimental): This is the same as the sitting condition, but participants will be asked to break their sitting time by standing close to their chair for 5 minutes, after 15 and 45 minutes of each hour following breakfast. The standing protocol will be repeated after lunch. Individuals will be asked to stand in the same position with no further instructions provided. In total, individuals will accumulate 12 bouts (60 minutes) of standing throughout the test period.
  Interventions: Behavioral: Standing
- Walking (Experimental): This is identical to the standing condition, but the breaks in sitting time will be punctuated with 5 minute bouts of light-intensity treadmill walking (equivalent to around 4.0km•h-1) rather than standing. In total, individuals will accumulate 12 bouts (60 minutes) of light-intensity activity throughout the test period. The light-intensity walking activity undertaken here replicates the low-grade ambulatory activity associated with everyday life.
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Sitting
  Arms: Sitting
Behavioral: Standing
  Arms: Standing
Behavioral: Walking
  Arms: Walking

SUMMARY:
The number of people diagnosed with Type 2 diabetes (T2DM) is increasing rapidly and about 2.9 million people in the UK currently have diabetes. There is increasing evidence suggesting that prolonged sedentary time may actually increase the risk of diabetes and other chronic diseases. Importantly, adults can meet public health guidelines on physical activity (150 minutes of moderate activity per week), but if they still sit for prolonged periods, their metabolic health is compromised. Going from sitting to standing and carrying out light-intensity activities (such as casual walking) may reduce diabetes risk. However, no one has investigated the effect of standing and walking on markers of cardio-metabolic markers in individuals with a high risk of T2DM. Therefore, the aim is to find out whether reducing the amount of time people spend sitting and replacing it with standing and light intensity activity (walking) reduces glucose, insulin and triglyceride levels, therefore reducing the risk of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary
* Overweight or obese (BMI>25kg/m2)
* Post menopausal
* Previous diagnosis of impaired glucose tolerance

Exclusion Criteria:

* Regular purposeful exercise (≥150 minutes of MVPA per week)
* Physical condition which limits full participation in the study
* Active psychotic illness or other significant illness which, in the view of the investigators, would prevent full participation
* Inability to communicate in spoken English
* Steroid use
* Known Type 2 Diabetes
* Pregnancy
* Male
* Currently taking hormone replacement medication.

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Glucose area under the curve | 0 weeks and 2 weeks
  Glucose area under the curve (AUC); Plasma glucose will be measured using a glucose oxidase method on the Beckman Auto Analyzer (Beckman, High Wycombe, UK). Glucose profile measurements will be undertaken in the same laboratory located within the Leicester Royal Infirmary.

SECONDARY OUTCOMES:
Insulin area under the curve | 0 weeks and 2 weeks
Triacylglycerol area under the curve | 0 weeks and 2 weeks
Lipoprotein lipase activity | 0 weeks and 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Melanie J Davies, MD, Principal Investigator — University of Leicester
Locations (1):
- Leicester Diabetes Centre, Leicester General Hospital, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Derived] Henson J, Davies MJ, Bodicoat DH, Edwardson CL, Gill JM, Stensel DJ, Tolfrey K, Dunstan DW, Khunti K, Yates T. Breaking Up Prolonged Sitting With Standing or Walking Attenuates the Postprandial Metabolic Response in Postmenopausal Women: A Randomized Acute Study. Diabetes Care. 2016 Jan;39(1):130-8. doi: 10.2337/dc15-1240. Epub 2015 Dec 1. PMID 26628415
- See also: Click here for more information about this study — http://www.ll.dlpa.bru.nihr.ac.uk